CLINICAL TRIAL: NCT05671042
Title: Neoadjuvant Chemotherapy in Upper Tract Urothelial Carcinoma : a Retrospective Multicentric Study.
Acronym: CNA TVES
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Other Study IDs: APHP220678
Record Dates: First submitted 2022-10-31; First posted 2023-01-04 (Actual); Last update posted 2023-01-04 (Actual); Status verified 2023-01

CONDITIONS: Upper Excretory Tract Tumors
MeSH Terms: interventions — Standard of Care

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients with Upper excretory tract tumors: Adult patient with Upper excretory tract tumors Neoadjuvant chemotherapy treatment received between 2010 and 2020.
  Interventions: Other: Patients with Upper excretory tract tumors

INTERVENTIONS:
Other: Patients with Upper excretory tract tumors — Standard of care for patients with Sezary Syndrome
  Other Names: Standard of care

SUMMARY:
Upper tract urothelial carcinoma incidence is about 1 /100000/year. These tumors are mostly diagnosed at an invasive stage and the standard treatment is a total nephroureterectomy.

In this population, indication of perioperative chemotherapy is still discussed. The benefit of platinum-based adjuvant chemotherapy was recently confirmed by the prospective trial POUT for pT2-T4 N0-3 M0 tumors with an improvement in recurrence-free survival of 51% in the chemotherapy arm.

However, in this situation, use of adjuvant Cisplatin-based chemotherapy may be limited by the deterioration of renal function due to renal surgery.

There are currently no recommendations on the place of neoadjuvant chemotherapy (NAC) with controversial results.

Moreover, the impact on renal function of the NAC-NUT treatment sequence has so far been little studied.

The aim of this study is to improve scientific knowledge about neoadjuvant chemotherapy in upper tract urothelial carcinoma eligible to a curative surgery. The investigators will evaluate the benefit of NAC on pathological response, overall survival and progression-free survival in a large multicentric cohort. In addition, the investigators will assess the impact of NAC on renal function at a distance from curative surgery will allow the evaluation of its specific toxicity.

ELIGIBILITY:
Inclusion Criteria:

1. Patients over 18 years of age
2. Male or female
3. Upper excretory tract tumors
4. Localized or locally advanced stage (N0 to N1)
5. Eligible for curative surgery
6. Have received neoadjuvant or primary chemotherapy
7. Neoadjuvant chemotherapy treatment received between 2010 and 2020.

Exclusion Criteria:

1. Patient's opposition to the research
2. UTUC not eligible for curative surgery
3. Locally advanced UTUC ≥ N2 and/or metastatic.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients with upper excretory tract tumors
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2023-01 (Estimated); Primary Completion 2023-05 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Pathological response rate | immediately after the end of chemotherapy treatment
  Pathological response rate on the surgical specimen after 4 to 6 cycles of chemotherapy (each cycle is 14 days or 21 days according to chemotherapy treatment).

SECONDARY OUTCOMES:
Progression free-survival | at one year
Progression free-survival | at 2 years
Progression free-survival | at 3 years
Progression free-survival | at 4 years
Radiological response rate | immediately after the end of chemotherapy treatment
  Radiological response rate before ablation surgery after 4-6 cycles of chemotherapy.
residual renal function assessed by creatinine clearance (mL/min) | at 3 months after curative surgery

IPD SHARING:
Plan to Share IPD: Undecided